CLINICAL TRIAL: NCT04773028
Title: The Role of Matrix Metalloproteinase 2 and 9 Enzymes in Developing Chronic Thromboembolic Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: AHMET ZENGIN (Other Government)
Responsible Party: Sponsor-Investigator, AHMET ZENGIN, medical doctor, Kartal Kosuyolu High Speciality Training and Research Hospital
Organization: Kartal Kosuyolu High Speciality Training and Research Hospital (Other Government)
Other Study IDs: 2020-071
Record Dates: First submitted 2021-02-19; First posted 2021-02-26 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples was teken from pulmonary endarterectomy material during the operation. This material is removed routinly this surgical procedure. At this studt any extra surgical procedure did not performed to participans.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PATİENT GROUP(GROUP 1): This group is the group that underwent pulmonary thromboendarterectomy due to chronic thromboembolic pulmonary hypertension.Sample was taken from the material extracted from this group during operation.
  Interventions: Other: matrix metalloproteinase enzymes 2 and 9
- CONTROL GROUP(GROUP 2): This group is the group that underwent lobectomy or pneumonectomy for another reason that the pulmonary artery is not affected. Patients operated for a reason other than chronic thromboembolic pulmonary hypertension and samples were taken from the intact pulmonary artery of the removed lung.
  Interventions: Other: matrix metalloproteinase enzymes 2 and 9

INTERVENTIONS:
Other: matrix metalloproteinase enzymes 2 and 9 — concentration of matrix metalloproteinase 2 and 9 enzymes

SUMMARY:
Chronic thromboembolic pulmonary hypertension is an occlusive disease in pulmonary artery.Matrix metalloproteinase enzymes play a substantial role of extracellular matrix remodeling. The clot formed in chronic thromboembolic pulmonary hypertension does not melt and turns into a fibrous state, it occludes the pulmonary artery.In this study, investigators aimed to investigate the role of matrix metalloproteinase enzymes in pulmonary arterial wall remodeling in patients with chronic thromboembolic pulmonary hypertension

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension is an occlusive disease in pulmonary artery. Only 4% of patients with acute pulmonary embolism develop chronic thromboembolic pulmonary hypertension and acute pulmonary embolism or deep vein thrombosis is reported in the anamnesis of 75% of those with chronic thromboembolic disease. Therefore, the etiology of the disease is not clear. Altought many studies are done, especially the role of inflamation is emhasised underlie the disease.

Matrix metalloproteinase enzymes play a substantial role of extracellular matrix remodeling. The clot formed in chronic thromboembolic pulmonary hypertension does not melt and turns into a fibrous state, it occludes the pulmonary artery.In this study, investigators aimed to investigate the role of matrix metalloproteinase enzymes in pulmonary arterial wall remodeling in patients with chronic thromboembolic pulmonary hypertension.

Matrix metalloprotinase enzymes are known to play a role in atherosclerosis. This research will investigate whether there is atherosclerosis together with inflamattion in the background of chronic thromboembolic hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Despite 3 months of anticoagulation therapy
* mean pulmonary arterial pressure > 20 mmHg
* pulmonary vasculary resistance > 3 wood
* pulmonary capillary wedge pressure < 15 mmHg
* perfusion defect in ventilation perfusion scintigraphy
* pulmonary angiography or computed tomography angiography showing pulmonary artery occlusive lesions

Exclusion Criteria:

* Patients undergoing pulmonary thromboendarterectomy concomitant coronary bypass, carotid endarterectomy, aortic valve, ascending aorta, mitral valve, tricuspid valve, pulmonary valve surgery
* Patients who have undergone surgical or percutaneous procedures due to atherosclerotic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population has chronic thromboembolic pulmonary hypertension and will be performed pulmonary thromboendarterectomy.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: mehmet yanartas, Study Director — kartal kosuyolu hıgh specıalty training and research hospital
Locations (1):
- Kartal Kosuyolu High Speciality Training and Research Hospital, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data used in the study will be kept closed to the use of other users.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PATİENT GROUP(GROUP 1) | CONTROL GROUP(GROUP 2)
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PATİENT GROUP(GROUP 1) | CONTROL GROUP(GROUP 2) | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 49.04 (10.8) | 57.8 (15.4) | 53.42 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 13 | 16 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 24 | 24 | 48
height [Mean (Standard Deviation); unit: cm] | 166.6 (10.2) | 166.7 (7.6) | 166.65 (8.9)
Weight [Mean (Standard Deviation); unit: kg] | 85.4 (14.2) | 73.5 (13.9) | 79.45 (14.05)

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Matrix Metalloproteinase 2 and 9 Enzymes
Description: Measurement the concentration of matrix metalloproteinase 2 and 9 enzymes by elisa and western blot techniques.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PATİENT GROUP(GROUP 1) | CONTROL GROUP(GROUP 2)
Number analyzed (Participants) | 24 | 24
ng/ml
  PRO MMP 2 | 89289.89 (84639.26) | 86548.72 (45312.33)
  ACTİVE MMP 2 | 205707.83 (388888.77) | 152911.57 (44400.16)
  MMP 9 | 88975.83 (94129.68) | 182029.76 (140527.87)
Statistical Analysis 1: Comparison: PATİENT GROUP(GROUP 1) vs CONTROL GROUP(GROUP 2); Test type: Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -93054

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/assessed
Description: Adverse Events were not monitored/assessed.
Arm/Group | PATİENT GROUP(GROUP 1) | CONTROL GROUP(GROUP 2)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT04773028/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT04773028/SAP_001.pdf